CLINICAL TRIAL: NCT01048996
Title: Genetic Variability and Biomarkers in Children With Acute Lung Injury
Acronym: BALI
Status: Withdrawn | Type: Observational
Why Stopped: PI has left institution
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); UCSF Benioff Children's Hospital Oakland (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 663
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; Genetic Variability; Plasma Biomarkers; Pediatrics
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 samples will be collected from each patient, one whole blood and three plasma samples will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non ALI/ARDS: Those patient who enrolled in the study but did not develop ALI or ARDS during their hospital course.
- ALI/ARDS: Those patients who enrolled in the study and developed ALI or ARDS during their hospital course.

SUMMARY:
Acute Lung Injury (ALI) and the more severe Acute Respiratory Distress Syndrome (ARDS) are a significant problem in Pediatric Intensive Care Units, affecting up to 16 of every 1000 children admitted to these units. These disorders carry with them high mortality rates as well as numerous long-term effects for the surviving children. As the effects of these diseases have significant social and economic ramifications for affected children and their families, research on the development of ALI/ARDS could significantly change how physicians understand the disease and treat patients.

There are a wide range of problems which make certain PICU patients more likely to develop either ALI or ARDS. This research aims to determine which of these children are at the greatest risk for ALI/ARDS by examining differences in plasma biomarkers and in DNA of a large number of PICU patients. We are hypothesizing that significant differences in the level of specific plasma biomarkers or in the frequency of specific DNA variants exist in children who develop ALI/ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive intubated pediatric patients (≥ 2 weeks of age and ≥ 42 weeks corrected gestational age and ≤ 18 years of age) supported on mechanical ventilation for acute pulmonary parenchymal disease enrolled in the RESTORE study.

Exclusion Criteria:

* Intubated and mechanically ventilated for immediate post-operative care and stabilization
* Cyanotic heart disease with unrepaired or palliated right to left intracardiac shunt
* History of single ventricle at any stage of repair
* Congenital diaphragmatic hernia or paralysis
* Primary pulmonary hypertension
* Critical airway (e.g., post laryngotracheal construction) or anatomical obstruction of the lower airway (e.g., mediastinal mass)
* Ventilator dependent (including noninvasive) on PICU admission (chronic assisted ventilation)
* Neuromuscular respiratory failure
* Spinal cord injury above the lumbar region
* Pain managed by patient controlled analgesia (PCA) or epidural catheter
* Family/medical team has decided not to provide full support (patient treatment considered futile)
* Enrolled in any other sedation clinical trial concurrently or within the last 30 days
* Known allergy to any of the study medications

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be recruited concurrently with subjects recruited for the "RESTORE" sedation study. All patients who have been admited to a Pediatric Intensive/Critical Care Unit and on mechanical ventilation will be screened for eligibility at the participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Development of ALI or ARDS | During PICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Michael Quasney, PhD, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States